CLINICAL TRIAL: NCT02739516
Title: Concomitant Administration of Follicle-stimulating Hormone at the Time of Human Chorionic Gonadotropin Trigger in Letrozole Stimulated Intrauterine Insemination Cycles in Women With Unexplained Infertility
Brief Title: Dual FSH/HCG Trigger in Letrozole Stimulated Intrauterine Insemination Cycles in Women With Unexplained Infertility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Walid Anwar Murad, Assistant Professor, Department of Obstetrics and Gynecology, Faculty of Medicine, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Benha 125
Record Dates: First submitted 2016-03-14; First posted 2016-04-15 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Chorionic Gonadotropin; Letrozole

ARMS (2):
- Control (Active Comparator): In letrozole stimulated cycle: On the day of ovulation trigger the patient received standard dose of Human chorionic gonadotropin (10,000 IU).
  Interventions: Drug: Human chorionic gonadotropin; Drug: Letrozole
- Study (Experimental): In letrozole stimulated cycle: On the day of ovulation trigger the patient received hCG 10000 IU plus FSH co-trigger (urofollitropin; Fostimon, IBSA, Bazel, Swiz; 75 IU amp) 150 IU injected once .
  Interventions: Drug: Human chorionic gonadotropin; Drug: FSH co-trigger; Drug: Letrozole

INTERVENTIONS:
Drug: Human chorionic gonadotropin — In letrozole stimulated cycle; Human chorionic gonadotropin ( hCG) 10000 IU was given intramuscular when the mean ovarian follicle diameter was ≥18 mm.
Drug: FSH co-trigger — In letrozole stimulated cycle; FSH (urofollitropin; Fostimon, IBSA, Bazel, Swiz; 75 IU amp) 150 IU injected once intramuscular when the mean ovarian follicle diameter was ≥18 mm.
  Arms: Study
Drug: Letrozole — Letrozole oral tablets (Femara 2.5 mg tablet; Novartis Pharma Services, Switzerland) 2.5 mg tab twice daily for 5 days from cycle day 3.

SUMMARY:
The objective of this study was to evaluate the outcome of follicle stimulating hormone (FSH) co-administration with human chorionic gonadotrophins trigger for women with unexplained infertility (UEI) and assigned for letrozole (LTZ) stimulated intrauterine insemination (IUI) cycles .

DETAILED DESCRIPTION:
This prospective randomized controlled study included 108 women with unexplained infertility recruited among those attending the Gynecology Outpatient Clinics of, Benha University Hospital, and private settings, Alkalubia, Egypt from Jun 2013 to Aug 2015. The study protocol was approved by the Local Ethics Committee and written informed consents were taken from both partners before starting of the study.

All women received the same regimen of ovarian stimulation using Letrozole (Femara; Novartis pharma AG, Basle, Switzerland) 2.5 mg tab twice daily for 5 days starting from cycle day 3. Transvaginal ultrasound scan (TVS) was performed daily from cycle day 9 and a total of 10,000 IU of hCG (Epifasi, EPICO) was administered to those in whom at least one ovarian follicle was ≥18 mm in size. On the day of hCG administration women were randomly categorized into two groups according to a computer generated random numerical table. Envelopes containing the allocation information were chosen sequentially by patient herself in presence of her husband. Group A received FSH (urofollitropin; Fostimon, IBSA, Bazel, Swiz; 75 IU amp) 150 IU injected once on day of hCG injection and group B received no FSH on day of hCG injection. Intrauterine insemination was performed 36 hours after HCG injection. Women in both groups received luteal phase support in the form of vaginal progesterone, (Prontogest 400 mg Vaginal Pessaries, IBSA) twice a day, starting from the day after IUI and continued till the eighth week, if the pregnancy test was positive.Two weeks later, quantitative ßhCG was estimated to diagnose chemical pregnancy. However, TVS was performed 4 weeks after positive pregnancy test to confirm clinical pregnancy by the presence of gestational sac with fetal echoes and pulsation and to exclude ectopic pregnancy. All women enrolled in the study underwent the study protocol for three consecutive cycles unless got pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility for more than 2 years
* Normal ovulation proved by midluteal serum progesterone level >5 ng/ml,
* Patent fallopian tubes confirmed by hysterosalpingography or laparoscopy
* Normal semen analysis according to the modified World Health Organization (WHO) criteria
* Normal hormonal profile (FSH, LH, prolactin and TSH) in the early follicular phase.

Exclusion Criteria:

* Other causes of infertility ( tubal factors, polycystic ovary syndrome (PCOS), endometriosis)
* Ovarian cysts,
* FSH >10 mIU/ml.
* Previous intrauterine insemination (IUI )cycles,
* Liver or kidney diseases,
* Hypersensitivity to the used medications.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate per cycle (PR/C) and per woman (PP/W) | Throughout the study completion; up to 3 months
  Achievement of clinical pregnancy defined as the presence of an intrauterine gestational sac with a pulsating fetal heart beat on ultrasound

SECONDARY OUTCOMES:
Frequency of ovarian hyperstimulation syndrome (OHSS) | Throughout the study completion; up to 3 months
  Number of participants developed ovarian hyperstimulation syndrome (OHSS) per all women received intervention
Multiple pregnancies | Throughout the study completion; up to 3 months
  Number of participants had multiple pregnancy per women achieved pregnancy .
The live birth rate per woman (LB/W). | Throughout the study completion; up to 2 year
  Number of live birth per women receiving intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Walid Anwar Murad, MD, Principal Investigator — Gynecology & Obstetric Department, Faculty of Medicine, Benha University